CLINICAL TRIAL: NCT04035109
Title: Anakinra as a Rescue Treatment for Nasal Allergen Challenge-induced Airway Inflammation
Brief Title: Anakinra as a Rescue Treatment for Allergic Inflammation
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study stopped due to COVID-19 pandemic.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 18-2650; 5R01HL135235 (NIH)
Record Dates: First submitted 2019-07-24; First posted 2019-07-29 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Asthma, Allergic
Keywords: asthma; nasal allergy; house dust mite; cat
MeSH Terms: conditions — Asthma | interventions — Interleukin 1 Receptor Antagonist Protein; Sodium Chloride; Antigens, Dermatophagoides

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Anakinra and matching saline placebo will be provided by the investigational drug service
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Anakinra (Period 1) then Placebo (Period 2) (Other): Subjects randomized to this arm will receive a single injection of anakinra 1 mg/kg (max dose of 100 mg) administered subcutaneously after their first allergen challenge (Period 1), followed by the matching saline placebo after their second allergen challenge (Period 2).
  Interventions: Drug: Anakinra; Drug: Preservative-free 0.9% sodium chloride (Placebo); Biological: House dust mite allergen; Biological: Cat hair allergen
- Placebo (Period 1) then Anakinra (Period 2) (Other): Subjects randomized to this arm will receive a single injection of saline placebo administered subcutaneously after their first allergen challenge (Period 1), followed by anakinra 1 mg/kg (max dose of 100 mg) administered subcutaneously after their second allergen challenge (Period 2).
  Interventions: Drug: Anakinra; Drug: Preservative-free 0.9% sodium chloride (Placebo); Biological: House dust mite allergen; Biological: Cat hair allergen

INTERVENTIONS:
Drug: Anakinra — A single 1mg/kg subcutaneous injection (up to 100mg) of anakinra will be administered after nasal allergen challenge.
  Other Names: Kineret
Drug: Preservative-free 0.9% sodium chloride (Placebo) — A single subcutaneous injection of sodium chloride (placebo) will be administered after nasal allergen challenge.
Biological: House dust mite allergen — Standardized house dust mite (Dermatophagoides farinae) allergen extract (provided by Greer Laboratories, Lenoir, NC). Participants who are sensitized to house dust mite (determined by skin prick testing) will undergo intranasal challenge with house dust mite allergen extract. All participants will undergo allergen challenge with a single allergen (house dust mite or cat hair).
  Other Names: Dermatophagoides farinae
Biological: Cat hair allergen — Standardized cat hair allergen extract (provided by Greer Laboratories, Lenoir, NC). Participants who are sensitized to cat hair (determined by skin prick testing) will undergo intranasal challenge with cat hair allergen extract. All participants will undergo allergen challenge with a single allergen (house dust mite or cat hair).
  Other Names: Felis catus

SUMMARY:
Participants with mild asthma who are sensitized to either house dust mite or cat hair allergen will undergo nasal instillation of the allergen to elicit nasal allergy symptoms. The participants will be treated in a cross-over fashion with either placebo (saline) or anakinra to determine if anakinra will reduce nasal airway eosinophil recruitment, eosinophil activation, release of inflammatory mediators, mucins, and gene expression changes in epithelial cells.

DETAILED DESCRIPTION:
Asthma is an increasingly common chronic illness with higher rates of hospitalization for exacerbation than many other chronic conditions. In 2009, total asthma costs in the U.S. were estimated at $56 billion per year, and over half the overall asthma-related costs were attributed to inpatient hospitalization. Allergen exposure and viral infection are among the most common triggers for asthma exacerbations. Exacerbations of allergic asthma are characterized by an early phase response, mediated by release of preformed mediators like histamine from mast cells, and a late phase response 3-7 hours later mediated by chemokines and cytokines, including IL-1beta (IL-1b), that attract leukocytes such as neutrophils and eosinophils to the airways, increase mucus production, trigger airway smooth muscle contraction, and result in airway constriction and airway hyper-reactivity.

While corticosteroids are considered a mainstay of treatment for asthma exacerbation regardless of the trigger, there are limitations to their effectiveness in the acute setting including the initial lag period of 4-6 hours or more before therapeutic effect and the concern for broad immune suppression. Corticosteroids are often ineffective in treating the neutrophilic component of airway inflammation seen with allergen-induced airway inflammation. Time to therapeutic benefit is key in preventing patient morbidity and mortality. Currently there is an urgent need for anti-inflammatory treatments that work quickly and effectively in acute asthma exacerbations.

The investigators propose that IL-1 blockade can achieve these ends and perhaps complement corticosteroid actions. Anakinra is an FDA-approved recombinant form of human IL-1 receptor antagonist (IL-1RA), a natural anti-inflammatory cytokine that competes with agonist binding to the IL-1 receptor, suppressing IL-1b and IL-1a signaling. Numerous murine and in vitro studies indicate that IL-1 signaling mediates key features of allergen-induced airway inflammation, including eosinophil recruitment and mucin production.

IL-1 receptor activity is important for eosinophil airway recruitment after allergen challenge through inducing endothelial cell adhesiveness and through increased mRNA expression of the eosinophil chemokine, eotaxin in pulmonary epithelial cells. IL-1 receptor type 1 (IL-1R1)-deficient mice demonstrate reduced allergic (eosinophilic) lung inflammation. Most pertinent to this project, anakinra treatment of wild type BALB/c mice prior to OVA challenge severely dampened airway eosinophil recruitment, cytokine responses, airway resistance and goblet cell numbers. In humans undergoing nasal allergen challenge, nasal secretions showed a biphasic pattern of IL-1b secretion that coincided with the early phase and late phase allergic responses. These data collectively suggest that IL-1 signaling is important in the allergic eosinophilic response and that anakinra has high potential to reduce eosinophilic inflammation.

Mucus accumulation is also a feature of allergen-induced inflammation and likely results from hypersecretion of mucus and failure of the mucociliary apparatus to effectively clear this mucus and airway debris. MUC5B and MUC5AC are the major secreted mucins in the human respiratory tract. IL-1b alone has been shown to induce increased epithelial cell mRNA expression of the mucin genes MUC5B and MUC5AC.

Anakinra is an ideal candidate to test as a rescue treatment for acute allergic inflammation due to its fast onset of action (reaching peak concentrations in 3-7 hours), and a short 4-6 hour half-life. Our objective is to determine if one treatment of anakinra mitigates a). eosinophil activation and recruitment and b) mucin secretion, after nasal allergen challenge, to ultimately assess if anakinra can mitigate key inflammatory features of asthma exacerbations. We expect that anakinra treatment will reduce nasal airway eosinophil recruitment, eosinophil activation, release of inflammatory mediators, mucins, and gene expression changes in epithelial cells after nasal allergen challenge based on pre-clinical data using anakinra with OVA challenge.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 18-45 years, inclusive
* Subjects will have mild asthma characterized by a Forced Expiratory Volume in 1 second (FEV1) of at least 75% of predicted and FEV1/FVC (Forced Vital Capacity) ratio of at least .60 (without use of bronchodilator medications for 12 hours), consistent with lung function of persons with mild episodic or mild persistent asthma. For the purpose of this protocol, an asthmatic individual will be defined as having a) positive methacholine challenge with a provocative concentration (PC) of methacholine producing a 20% fall in FEV1 (Provocative Concentration to decrease FEV1 by 20% (PC20) methacholine) with less than or equal to 10 mg/ml; OR b) physician-diagnosed asthma.
* OR non-asthmatic individuals with allergic rhinitis
* Allergic sensitization to house dust mite (Dermatophagoides farinae) OR cat (Felis catus) as confirmed by positive immediate skin prick test response (identified previously on a general screening visit)
* Negative pregnancy test for females who are not status post hysterectomy with oophorectomy or who have not been amenorrheic for 12 months or more.
* Ability to withhold antihistamine medications for one week prior to baseline and allergen challenge visits.
* Negative quantiferon gold TB test positive tuberculosis (TB) test is a contraindication to anakinra injection). A negative TB test within the past year (either tuberculin skin test (TST) with less than 5 mm induration or negative quantiferon TB Gold) is also acceptable.
* Subjects must be able and willing to give informed consent.

Exclusion Criteria:

* Any chronic medical condition considered by the PI as a contraindication to participation in the study including significant cardiovascular disease, diabetes, chronic renal disease, chronic thyroid disease, history of chronic infections or immunodeficiency.
* Pregnancy or nursing a baby.
* History of latex allergy/sensitivity
* Allergy/sensitivity to anakinra or its formulation
* Physician directed emergency treatment for an asthma exacerbation within the preceding 12 months.
* Exacerbation of asthma more than 2x/week which could be characteristics of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma.
* Daily requirements for albuterol due to asthma symptoms (cough, wheeze, chest tightness) which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma (not to include prophylactic use of albuterol prior to exercise).
* Viral upper respiratory tract infection within 4 weeks of challenge.
* Any acute infection requiring antibiotics within 4 weeks of exposure or fever of unknown origin within 4 weeks of challenge.
* Severe asthma
* Mental illness or history of drug or alcohol abuse that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements.
* Cigarette smoking >1 pack per month
* Nighttime symptoms of cough or wheeze greater than 1x/week at baseline (not during a clearly recognized viral induced asthma exacerbation) which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma.
* Allergy/sensitivity to study drugs or their formulations
* Known hypersensitivity to methacholine or to other parasympathomimetic agents
* History of intubation for asthma
* Unwillingness to limit coffee, tea, cola drinks, chocolate, or other foods containing caffeine after midnight on the days that methacholine challenge testing and nasal allergen challenge is to be performed.
* Unwillingness to use reliable contraception if sexually active (IUD, birth control pills/patch).

Usage of the following medications:

* Use of systemic steroid therapy within the preceding 12 months for an asthma exacerbation. All use of systemic steroids in the last year will be reviewed by a study physician.
* Subjects who are prescribed daily inhaled corticosteroids, cromolyn, or leukotriene inhibitors (Montelukast or Zafirlukast) will be required to discontinue these medications at least 4 weeks prior to their screening visit.
* Use of daily theophylline within the past month.
* Daily requirement for albuterol due to asthma symptoms (cough, wheeze, chest tightness) which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma. (Not to include prophylactic use of albuterol prior to exercise).
* Use of any immunosuppressant therapy within the preceding 12 months will be reviewed by the study physician.
* Use of any immunomodulatory therapy within the preceding 12 months.
* Use of beta blocking medications
* Antihistamines in the 5 days prior to allergen challenge
* Routine use of non-steroidal anti-inflammatory drugs (NSAIDs), including aspirin.

Physical/laboratory indications:

* Abnormalities on lung auscultation
* Temperature >37.8 C
* Oxygen saturation of <94%
* Systolic BP>150 mmHg or <90 mmHg or diastolic BP>90 mmHg or <60 mmHg
* Absolute neutrophil count (ANC) <1.4 x 109/L

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Change in eosinophils per milliliter of Nasal Lavage Fluid (NLF) | 6 hours post-allergen challenge versus pre-allergen challenge
  Allergen-induced eosinophil recruitment will be measured by measuring eosinophil content of fluid obtained from lavage of the nares, comparing pre-challenge lavage samples to samples obtained 6 hours after allergen challenge

SECONDARY OUTCOMES:
Change in neutrophils per milliliter of NLF | 6 hours post-allergen challenge versus pre-allergen challenge
  Allergen-induced neutrophil recruitment will be measured by measuring neutrophil content of fluid obtained from lavage of the nares, comparing pre-challenge lavage samples to samples obtained 6 hours after allergen challenge
Change in inflammatory cytokines in nasal epithelial lining fluid (ELF) | 6 hours post-allergen challenge versus pre-allergen challenge
  Allergen-induced changes in inflammatory cytokines will be measured by measuring concentrations of these products in nasal epithelial lining fluid obtained through use of absorbent paper strips placed into the nares, comparing pre-challenge samples to samples obtained 6 hours after allergen challenge
Change in secreted mucin, MUC5AC, in NLF | 6 hours post-allergen challenge versus pre-allergen challenge
  Allergen-induced changes in MUC5AC in fluid obtained by lavage of the nares, comparing pre-challenge samples to samples obtained 6 hours after allergen challenge
Change in secreted mucin, MUC5B, in NLF | 6 hours post-allergen challenge versus pre-allergen challenge
  Allergen-induced changes in MUC5B in fluid obtained by lavage of the nares, comparing pre-challenge samples to samples obtained 6 hours after allergen challenge
Change in Nonspecific bronchial reactivity (NSBR) | 24 hours post-allergen challenge versus pre-allergen challenge
  NSBR will be assessed before and 24 hours after allergen challenge using methacholine challenge, which measures the responsiveness of the airways to a standard cholinergic bronchoconstriction agent (non-specific airway reactivity).
Change in Eosinophilic cationic protein (ECP) in nasal ELF | 6 hours post-allergen challenge versus pre-allergen challenge
  Allergen-induced changes in ECP, a marker of eosinophil activation, will be measured by measuring concentrations of ECP in nasal ELF obtained through use of absorbent paper strips placed into the nares, comparing pre-challenge samples to samples obtained 6 hours after allergen challenge

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Hernandez, Principal Investigator — Associate Professor of Pediatrics

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 9 to 36 months following publication
Access Criteria: Approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and execution of a data use/sharing agreement with UNC.